CLINICAL TRIAL: NCT06684418
Title: Artificial Intelligence-based Model for the Prediction of Occult Lymph Node Metastasis and Improvement of Clinical Decision-making in Non-small Cell Lung Cancer: A Multicenter, Prospective, Observational Study
Brief Title: Artificial Intelligence-based Model for the Prediction of Occult Lymph Node Metastasis and Improvement of Clinical Decision-making in Non-small Cell Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhengfei Zhu, Professor, Fudan University
Other Study IDs: OLNM-AI
Record Dates: First submitted 2024-11-11; First posted 2024-11-12 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: NSCLC (Non-small Cell Lung Cancer); Artificial Intelligence (AI); Lymphnode Metastasis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 50 patients will be selected to analyze the histopathology of the lesions and explore the relevant characteristics. RNA sequencing and multicolor fluorescence staining will be performed to explore differential genes and enriched signaling pathways. The tumor immune microenvironment will also be analyzed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective Cohort: Enrolling about 5,000 early-stage NSCLC patients from January 2018 to June 2024 across 25 centers in China, data including chest CT scans and clinicopathological parameters will be used to train and validate the AI model. Patients will be divided into "high-risk" and "low-risk" groups based on the model's risk score, and clinical benefits of treatments like lymph node dissection, adjuvant therapy, and SBRT will be analyzed.
  Interventions: Diagnostic Test: chest enhanced CT
- Prospective Cohort: Enrolling 1,000 patients from November 2024 to October 2025, this cohort will prospectively validate the AI model's performance and explore the biological basis of metastasis by analyzing pathological tissues, RNA sequencing, and tumor immune microenvironment characteristics.
  Interventions: Diagnostic Test: chest enhanced CT

INTERVENTIONS:
Diagnostic Test: chest enhanced CT — This is an observational study and patients will receive routine clinical treatment according to the corresponding guidelines. We will collect the enrolled patient's chest enhanced CT and clinicopathological parameters.

SUMMARY:
This nationwide, multicenter observational study aims to develop and validate a multimodal artificial intelligence (AI) model for detecting occult lymph node metastasis in early-stage non-small cell lung cancer (NSCLC) patients. Despite advances in lymph node staging, 12.9%-39.3% of occult nodal metastasis cases remain undetected preoperatively, affecting treatment decisions. This study will use deep learning to extract imaging features of occult metastasis and combine them with clinical data to build an AI model for risk prediction. This study will provide insights into the feasibility of AI-driven detection of occult metastasis, supporting clinical decision-making and potentially revealing underlying biological mechanisms of lymph node metastasis in NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed non-small cell lung cancer;
* Clinical stage I (AJCC, 8th edition, 2017);
* Age≥18 years old;
* KPS score≥70;
* Patients who have undergone primary NSCLC radical surgery or SBRT treatment;
* Complete systemic lesion imaging assessment before primary NSCLC radical surgery or SBRT treatment (Note: Tumor size ≥ 3 cm or centrally located tumor requires PET/CT and/or invasive mediastinal staging);
* Patients willing to cooperate with the follow-up after primary NSCLC radical surgery;
* informed consent of the patient.

Exclusion Criteria:

* Poor quality of computed tomography imaging;
* Baseline imaging shows pure ground-glass nodules (GGO);
* Uncontrolled epilepsy, central nervous system disease, or history of mental disorders, judged by the researcher to potentially interfere with the signing of the informed consent form or affect patient compliance.;
* Loss to follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Early-stage NSCLC receiving curative treatment (surgery or SBRT).
Sampling Method: Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival (RFS) | 1 year
  The time from surgical treatment or SBRT to disease recurrence or death. Patients who were still not progressing at the time of analysis will have the date of their last contact as the cutoff date.

SECONDARY OUTCOMES:
Overall Survival (OS) | 1 year
  The time from the surgery or SBRT until death from any cause. Patients who are still alive at the time of analysis will have their last contact date used as the cutoff date.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan university Shanghai Cancer Center, Shanghai, China